CLINICAL TRIAL: NCT06083805
Title: Reliability and Validity of the Turkish Version of the Manual Ability Index in Elderly Population
Brief Title: Manual Ability Index in Elderly Population
Status: Completed | Type: Observational
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Menekse Safak, Res. Assist., Suleyman Demirel University
Other Study IDs: MS2023/03
Record Dates: First submitted 2023-09-28; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Elderly
Keywords: Elderly; Manual Ability Index; Reliability; Validity; Turkish version

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to conduct a Turkish validity and reliability study of the hand ability scale in the elderly population. Thus, the psychometric properties of the scale, which evaluates hand use in daily life activities in detail and functionally, will be determined in the elderly and an alternative method will be created to evaluate hand functions in the elderly.The sample of the study consists of 220 elderly individuals aged 65 and over residing in the city center of Isparta. Two independent native Turkish translators performed forward translation. To ensure clinical consistency, it was sent to an expert committee of seven expert physiotherapists, 2 neurologists, 1 gerontologist, and 2 translators with no medical or clinical background to reveal vague concepts in the original questionnaire. A single consequent Turkish translation was formed from the combination of the two translations The Turkish scale was translated back into English by two English-native speakers who speak Turkish fluently, and the English version of the scale was compared to the original. A group of experts authorized the final version of the document in Turkish, which was back ward translation. Translators reviewed the translations and compared certain inconsistencies.

DETAILED DESCRIPTION:
Aging is a complex multifactorial process, the basic mechanism of which is not fully elucidated and leads to deterioration of biological functions.It is stated that the loss of hand function seen in the elderly leads to poor performance in activities of daily living and recreational activities. For this reason, performance measurements in the elderly should include hand function measurement and aim to measure the adequacy and participation of the functions that the elderly person frequently uses in daily life activities. Scales applied to evaluate hand function are generally performance-based. The hand ability scale is among the scales that evaluate hand functions. The scale is used in the subjective evaluation of upper extremity functions and many parameters related to daily living activities in neurological and musculoskeletal problems.Healthy volunteers over the age of 65 were reached from various centers in Isparta, especially the applications made through the announcements on the bulletin boards on the Süleyman Demirel University campus. Each participant was informed about the content of the study, and the volunteers read and signed informed consent forms. Before the formal questionnaire, the pre-final Turkish version of the questionnaire was used for a pilot test. The Turkish translation was primarily applied to five participants for the detection of unintelligible questions or words. Turkish translation was applied to five participants in order to determine the questions or words that were not understood. Investigators asked the participants the following questions: "Is there a question you don't understand?" "Are there any words you don't like?" Since the participants did not have any problems, no changes were made in the questionnaire and the final Turkish version of the MAM (MAM-T) was provided.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older,
* Being literate,
* Volunteering to participate in the research,
* It means getting a score of 24 or above when the Standardized Mini Mental Test Score is applied.

Exclusion Criteria:

* Having a condition that prevents them from performing daily life activities,
* Having serious vision and hearing loss,
* Having any neurological, orthopedic or rheumatological comorbidities that may affect hand functions, such as diagnosed stroke, carpal tunnel, lateral epicondylitis,
* Having a diagnosed psychiatric disorder,
* Lack of cooperation,
* Being in the recovery period of an acute illness.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The sample of the study consists of 220 elderly individuals aged 65 and over residing in the city center of Isparta. The GPower 3.1 program was used to determine the sample size of the study. When the effect size was calculated according to the number of samples taken from a similar study, a rate of 0.24/0.47 was found (8). However, in our study, by choosing the binomial test in the GPower program; after the calculation with an effect size of 0.24 and a power of 95%, it was determined that the sample size should be at least 190 elderly people. In the literature, it is stated that when determining the sample size for factor analysis, an acceptable sample size of 4:1 or 5:1 per item will be sufficient (9).
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Manuel Ability Measure | 2023
  The Manual Ability Measure-36 (MAM-36) is a 36-item scale that assesses perceived ease or difficulty in performing daily activities (e.g., eating, dressing, buttoning clothes) using one's hands, regardless of which hand is used and excluding the use of assistive equipment. It is scored between 0 and 4 points according to the Likert scale.

SECONDARY OUTCOMES:
Duruöz Hand Index | 2023
  The Duruöz Hand Index (DHI) was first developed in 1996 for the assessment of hand functions in patients with rheumatoid arthritis; It is a valuable test with proven validity and reliability in many diseases related to the upper extremity. The test consists of 18 questions and is presented by separating daily life functions, does not require additional training and equipment for the test, and is a simple, useful and reliable test that takes approximately 3-5 minutes to apply. Answers are given on a Likert scale, and a lower score indicates better functional status.
Mini Mental State Test | 2023
  Mini Mental State Test (MMDT) will be used to evaluate the cognitive functions of individuals. The test, which is gathered under 6 main headings as orientation, recording memory, attention and calculation, recall and language, is evaluated over a total of 30 points. A value of 24 is accepted as the threshold value, and a decrease in this value indicates deterioration in cognitive functions. The validity and reliability study of the test was performed by Güngen et al.

CONTACTS AND LOCATIONS:
Overall Officials: Adnan KARAİBRAHİMOĞLU, Assist. Prof., Study Director — Suleyman Demirel University; Menekşe ŞAFAK, Res. Assist., Principal Investigator — Suleyman Demirel University; Mert USTA, Res. Assist., Principal Investigator — Suleyman Demirel University; Ferdi BAŞKURT, Prof. Dr., Principal Investigator — Suleyman Demirel University; Zeliha BAŞKURT, Prof. Dr., Principal Investigator — Suleyman Demirel University
Locations (1):
- Menekşe ŞAFAK, Isparta, Merkez, Turkey (Türkiye)